CLINICAL TRIAL: NCT00403819
Title: A Phase III Multi-Centre Placebo-Controlled Crossover Study Followed by an Open Label Post-Study Follow-up to Examine the Efficacy and Safety of Movicol in the Treatment of Chronic Constipation in Children
Brief Title: Study to Examine the Efficacy and Safety of Movicol in the Treatment of Chronic Constipation in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Norgine (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2000/01
Record Dates: First submitted 2006-11-24; First posted 2006-11-27 (Estimated); Last update posted 2006-11-28 (Estimated); Status verified 2006-11

CONDITIONS: Chronic Constipation

INTERVENTIONS:
Drug: Polyethylene glycol 3350 Na bicarbonate NaCl KCl (Movicol)

SUMMARY:
A phase III, multi-centre, double blind, placebo controlled, crossover study, followed by an open label post study follow-up, to assess the efficacy and safety of Movicol in the treatment of chronic constipation in children

DETAILED DESCRIPTION:
After a baseline period of 1 (one) week, subjects who had met the inclusion criteria were entered into the treatment phase of the study. Patients were randomised to receive either Movicol or matching Placebo for two (2) weeks. Following the treatment phase, patients underwent a two (2)-week placebo washout period prior to crossing over to receive the alternative treatment e.g. those patients who took Movicol were given the matching Placebo or vice versa on completion of the washout period for two (2) weeks.

On completion of the double blind treatment phase, patients were given the option to participate in the eight (8) week open label post study follow-up. Patients who participated in the post study follow-up received Movicol.

ELIGIBILITY:
Inclusion Criteria:

Male and female patients of any ethnic origin will be eligible to participate in the study if all of the following criteria are fulfilled.

* informed consent having been obtained from the patient's parent or guardian and assent from the child if they are capable of understanding the study
* aged 24 months - 11 years
* experiencing constipation as defined as:

  * ≤2 complete bowel movements per week, and at least one of the following:

    * pain on defaecation on ≥1 in 4 days
    * 1/4 or more of bowel movements with straining
    * 1/4 or more of bowel movements with hard or lumpy stools
* patients in whom these symptoms have been present for ≥3 months
* available to complete the study and able to comply with requirements and restrictions listed in the patient's/parent's information documents.

Exclusion Criteria:

Patients will not be eligible to participate in the study if any of the following conditions apply:

* faecal impaction or history of faecal impaction
* history of intestinal perforation or constipation
* paralytic ileus
* toxic megacolon
* Hirschsprungs disease
* severe inflammatory conditions of the intestinal tract
* severe gastro-oesophageal reflux - that which is complicated by anaemia, haematemesis, respiratory aspiration, failure to thrive or other recognised complications of gastro-oesophageal reflux
* patients currently receiving over 0.5mg/kg/day of senna or over 1/2 sachet of sodium picosulphate per day for children <6 years and over 1 sachet sodium picosulphate per day for children > 6 years (i.e. high doses of stimulant laxatives)
* any other significant medical condition that in the investigator's opinion would effect their suitability for entry into the study
* patients who have previously received Movicol or previously participated in the study
* known hypersensitivity to polyethylene (PEG) 3350 or any of the constituents of Movicol
* patients with diabetes as the placebo to be used in this study is sucrose
* patients who have received any investigational drug in the last 3 months
* patients and/or parents who the investigator thinks could not comply with the requirements of the protocol for any reason (particularly in relation to reliable completion of diary cards)

Ages: 24 Months to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60
Dates: Start 2002-04; Study Completion 2003-04

PRIMARY OUTCOMES:
Mean number of complete defaecations per week in each treatment period

SECONDARY OUTCOMES:
Mean total number of defaecations (complete plus incomplete) per week in each treatment period
Pain on defaecation
Straining on defaecation
Abdominal pain
Faecal incontinence
Stool consistency

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Thomson, MD, Principal Investigator — Royal Free Hospital NHS Foundation Trust
Locations (6):
- United Kingdom (6):
  - Aberdeen Children's Hospital, Aberdeen
  - University Hospital of Wales, Children's Hospital, North Ward, Cardiff
  - Royal Hospital for Sick Children, University Hospitals NHS Trust, Edinburgh
  - Leicester Royal Infirmary, Leicester
  - Royal Free Hospital, London
  - New Cross Hospital, Royal Wolverhampton Hospitals NHS Trust, Wolverhampton

REFERENCES:
- [Background] Issenman RM, Hewson S, Pirhonen D, Taylor W, Tirosh A. Are chronic digestive complaints the result of abnormal dietary patterns? Diet and digestive complaints in children at 22 and 40 months of age. Am J Dis Child. 1987 Jun;141(6):679-82. doi: 10.1001/archpedi.1987.04460060095043. PMID 3578195
- [Background] Hatch TF. Encopresis and constipation in children. Pediatr Clin North Am. 1988 Apr;35(2):257-80. doi: 10.1016/s0031-3955(16)36431-8. PMID 3278282
- [Background] Loening-Baucke V. Constipation in early childhood: patient characteristics, treatment, and longterm follow up. Gut. 1993 Oct;34(10):1400-4. doi: 10.1136/gut.34.10.1400. PMID 8244110
- [Background] Benninga MA, Buller HA, Heymans HS, Tytgat GN, Taminiau JA. Is encopresis always the result of constipation? Arch Dis Child. 1994 Sep;71(3):186-93. doi: 10.1136/adc.71.3.186. PMID 7979489
- [Background] Benninga MA, Buller HA, Tytgat GN, Akkermans LM, Bossuyt PM, Taminiau JA. Colonic transit time in constipated children: does pediatric slow-transit constipation exist? J Pediatr Gastroenterol Nutr. 1996 Oct;23(3):241-51. doi: 10.1097/00005176-199610000-00007. PMID 8890073
- [Background] Culbert P, Gillett H, Ferguson A. Highly effective new oral therapy for faecal impaction. Br J Gen Pract. 1998 Sep;48(434):1599-600. PMID 9830188
- [Result] Thomson M, Jenkins H, et al. A Placebo Controlled Crossover Study of Movicol in the Treatment of Childhood Constipation. J Pediatr Gastroenterol Nutr 2004;39(1):S16 [abstract]